CLINICAL TRIAL: NCT01939080
Title: Exercise Training in Patients With Cardiovascular Risk: Predictability of Aortic Compliance Normalization
Brief Title: Variation of Aortic Compliance Related to Exercise Training With or Without Supervised Sessions
Acronym: ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12/B/01; 2012-A00359-34 (Other: AFSSAPS)
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Cardiovascular Disease
Keywords: moderate risk; high risk
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical supervision (Active Comparator): Exercise training with supervised sessions Classics training
  Interventions: Procedure: Exercise training with supervised sessions
- No medical supervision (Active Comparator): Exercise training without supervised sessions Classics training
  Interventions: Procedure: Exercise training with supervised sessions

INTERVENTIONS:
Procedure: Exercise training with supervised sessions

SUMMARY:
Many conditions and cardiovascular diseases (including stroke) are better managed with regular exercise training. The expected effects are partial reversal of adverse effects on heart and blood vessel structure and function, improved glycemic, tension and weight control.

Physiologically, the aorta maintains low left ventricular after-load, promotes optimal sub-endocardial coronary blood flow, and transforms pulsatile into laminar blood flow. Increased aortic stiffness may ultimately contribute to left ventricular dysfunction. Regular exercise training is likely to decrease the pulse wave velocity (a measure of the aortic compliance). Some subjects seem more responsive than others, and they may not expect the same benefit of exercise training. To the best of our knowledge, this has not been explained yet.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 50-69 years, with moderate or high cardiovascular risk

Exclusion Criteria:

* any physical or medical problem liable to limit the patient' ability to perform the cardiopulmonary exercise testing or the exercise training in safe conditions.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | With or without the exercise training

SECONDARY OUTCOMES:
Heart rate variability | within 12 weeks after exercise training

CONTACTS AND LOCATIONS:
Locations (2):
- CHU de Pointe à Pitre, Pointe-à-Pitre, Guadeloupe
- CHU de Fort de France, Fort-de-France, Martinique